CLINICAL TRIAL: NCT01415635
Title: Positive Effect of Fortified Hospital Food on Nutritional Intake in Patients at Nutritional Risk. A Randomized Controlled Trial.
Brief Title: Fortified Hospital Food as Nutritional Support
Acronym: DHH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-1-2011-048
Record Dates: First submitted 2011-07-19; First posted 2011-08-12 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Malnutrition
Keywords: Nutritional risk, Hospital food, Nutritional Intervention
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nutritional intervention (Experimental): The study will compare standard nutritional care (control group) with tailored nutritional care (the possibility to order small energy and protein-enriched dishes called "Delights of Herlev Hospital")(intervention group).
  Interventions: Dietary Supplement: Nutritional intervention using

INTERVENTIONS:
Dietary Supplement: Nutritional intervention using — The study is af 12 week randomized clinical trail with inclusion of 96 patients at nutritional risk, according to the NRS-2002 system. The intervention group is is given a tailored nutritional care(the possibility to order small energy and protein-enriched dishes called "Delights of Herlev Hospital").

SUMMARY:
Background:

The investigators have previously documented that patients at nutritional risk lack sufficient energy and protein intake. In 2009 the investigators conducted a non-randomized historically controlled intervention study of 40 patients at nutritional risk. The study indicated that a tailored food concept increased nutritional intake in this patient group.

The objective of the current study is therefore to investigate these findings in a randomized clinical trial. Our target is for 75% of patients in the intervention group to reach 75% of their energy and protein requirements.

Methods:

The study will compare standard nutritional care (control group) with tailored nutritional care (the possibility to order small energy and protein-enriched dishes called "Delights of Herlev Hospital"). 96 patients at nutritional risk, according to the NRS-2002 criteria, will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* patients at nutritional risk, according to the NRS-2002 system
* patients must be able to understand the information and be able to give a written informed consent (sufficient cognitive functioning)
* well-functioning gastrointestinal tract
* anticipated length of hospitalization of more than 3 days

Exclusion Criteria:

* terminal patients
* dysphagia
* food allergy or intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was the percentage of patients reaching >75% of their protein and energy requirements. | Energy and protein intake will be calculated on an average of 3 and up to 7 days of dietary. Number of days of food intake recording depends on how long the patient is hospitalized.
  The patients energy requirement will be estimated both from the factorial method and by Harris and Benedicts formula. Protein requirement will be 18E% of the energy requirement.
  Recording of the dietary intake will be carried out on a daily basis over a periode of minimum 3 days and maxium 7 days

SECONDARY OUTCOMES:
handgrip strength | at day 3, 5 and 7
  Handgrip strength (HGS)will be measured with a Jamar Digital Hand Dynanometer. HGS will only be measured in the right hand because the right hand i significantly stronger in right-handed subjects and there is no significant difference between the two sides in left-handed subjects. Subjects will be encouraged to perform maximal contractions three times with a 15-s interval and the average value will be recorded.
average daily energy and protein intake | Patient und energy and protein intake will be followed during hospitalization from enrollment in the study and until discharge or up to 7 days
Use of tube feeding | The patients use of tube feeding will be followed from enrollment in the study and until discharge, an expected average of 9 days.
  Use of tube feeding will be registrated (yes or no and amount (ml.)
use of parenteral nutrition | The patients use of parenteral nutrition will be followed from enrollment in the study and until discharge, an expected average of 9 days.
  Registration of use of parenteral nutrition (yes or no). If yes how much (ml.).
length of stay | an expected average of 9 days.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Munk, MSc., Study Director — Herlev University Hospital, Denmark
Locations (1):
- Herlev University Hospital, Herlev, Copenhagen, Denmark

REFERENCES:
- [Background] Hansen MF, Nielsen MA, Biltz C, Seidelin W, Almdal T. Catering in a large hospital--does serving from a buffet system meet the patients' needs? Clin Nutr. 2008 Aug;27(4):666-9. doi: 10.1016/j.clnu.2008.05.004. Epub 2008 Jul 14. PMID 18621450